CLINICAL TRIAL: NCT00368147
Title: Access Creation for Hemodialysis: Potential Contribution to Left Ventricular Remodelling
Brief Title: Access Creation for Hemodialysis: Association With Structural Changes of the Heart
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Kidney Foundation of Canada (Other)
Responsible Party: Deborah Zimmerman, Kidney Research Centre
Other Study IDs: 2002027-01H
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Arteriovenous Fistula; Arteriovenous Graft; Left Ventricular Hypertrophy; Brain Natriuretic Peptide
Keywords: Hemodialysis; Arteriovenous Fistula; Arteriovenous Graft; Left Ventricular Hypertrophy; Brain Natriuretic Peptide
MeSH Terms: conditions — Arteriovenous Fistula; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the creation of a fistula or a graft plays a role in the development of heart disease for patients undergoing hemodialysis

DETAILED DESCRIPTION:
Patients with end stage renal disease are at 18-20 times greater risk of dying from cardiovascular disease as the general population. Both traditional and non-traditional cardiovascular risk factors are thought to be important. Of the non-tradtional cardiovascular risk factors, creation of an arteriovenous fistula or graft for the purposes of a blood access for hemodialysis may contribute to an elevation in BNP and left ventricular hypertrophy - both factors that have been associated with an increased risk of mortality Prior to access creation and at one month and one year post access creation - samples for BNP will be collected Prior to access creation and at one year post access creation - echocardiography will be performed

ELIGIBILITY:
Inclusion Criteria: 1)Hemodialysis 2)high risk for heart failure (DM, age>50, and/or systolic dysfunction) 3) first arteriovenous fistula/graft 4) informed consent 5) technically adequate echocardiogram 6) stable hgb(>100) 7) stable mineral metabolism (normal calcium, phosphate <2.1mmol/L, PTH>50pmol/L)

Exclusion Criteria: 1)Expected survival <1 year 2) Expected to get a living donor transplant in one year 3)primary access failure 4) ARF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2002-04; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Zimmerman, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- University Heatlh Network, Toronto, Ontario, Canada